CLINICAL TRIAL: NCT02625142
Title: Engaging Families in Bedside Rounds to Promote Pediatric Patient Safety
Brief Title: Family-Centered Rounds Checklist Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: M-2010-1277; HS018680 (Other Grant/Funding Number: AHRQ)
Record Dates: First submitted 2015-11-02; First posted 2015-12-09 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Child, Hospitalized; Delivery of Health Care; Morning Rounds
Keywords: Morning Rounds; Patient-centered Care; Hospital Medicine; Pediatrics; Hospitals, Pediatric

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-centered rounds checklist (Experimental): During the "post-intervention" period, health care team members on two pediatric inpatient services received the Family-centered Rounds Checklist tool, as well as training in how to use the checklist in the delivery of effective family-centered rounds
  Interventions: Other: Family-centered rounds checklist tool
- Usual care (No Intervention): Two pediatric inpatient services were not provided the Family-centered rounds checklist tool, and delivered morning rounds in their usual manner. These services served as a control.

INTERVENTIONS:
Other: Family-centered rounds checklist tool — A printed checklist containing 9 key tasks associated with effective delivery of family-centered rounds. A previously-identified member of each rounding team was responsible for holding the printed checklist during morning rounds. Team members were trained the in the use of this checklist prior to the post-intervention period, and a brief refresher training was conducted mid-way through the period.
  Arms: Family-centered rounds checklist

SUMMARY:
The goal of this study is to develop, implement, and evaluate the effectiveness of an intervention designed to facilitate family engagement during bedside rounds at a children's hospital. The intervention consists of a "checklist" of key behaviors associated with the delivery of quality family-centered rounds, as well as training in the use of the checklist tool. In a pre-post controlled design, two hospital services will be randomized to use the checklist while two others will be randomized to usual care. The intervention is expected to increase to the performance of key checklist behaviors, family engagement, and family perceptions of patient safety.

DETAILED DESCRIPTION:
Family engagement in children's healthcare encounters has been suggested as a means to improve safety. To engage families in care, the recommended practice is to conduct rounds at the child's bedside with the family present (family-centered rounds). Family-centered rounds strive to engage families in (1) a relationship with care providers, (2) exchange of information for decision making, and (3) deliberation about decisions. Bedside rounds represent a consistent venue to engage families in the care of hospitalized children, yet no studies have systematically identified and examined the barriers and facilitators of family engagement during rounds as a means to improve safety.

ELIGIBILITY:
Inclusion Criteria:

* Admitted as an inpatient on the pediatric hospitalist service, pulmonary service, or hematology/oncology service, during the study period.

Exclusion Criteria:

* Stigmatizing/sensitive reason for hospitalization (e.g., suspected non-accidental trauma or mental health concerns)
* New cancer diagnosis
* Parent(s) unable to speak or read English
* Parent(s) unavailable to consent (absent or sleeping during recruitment visits)
* Already participated in the study during a prior inpatient admission

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 340 (Actual)
Dates: Start 2010-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Parent perceptions of hospital safety climate | Change between baseline (inpatient admission) and study completion (discharge from hospital, an average of 6 days)
  Children's Hospital Safety Climate survey
Family engagement in rounds | Every family-centered morning round that occurred during the patient's hospital stay through study completion, an average of 6 days
  Video data was collected for every morning round over the course of the patient's hospital stay. These videos were coded for measures of family engagement in rounds using established and validated coding systems (e.g. RIAS).

SECONDARY OUTCOMES:
Checklist item performance | Every family-centered morning round that occurred during the patient's hospital stay through study completion, an average of 6 days
  Assessment of how many key checklist elements were performed during each family-centered round (coded from video recordings of each round).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth D Cox, MD PhD, Principal Investigator — Dept. of Pediatrics, School of Medicine and Public Health, UW-Madison
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health; American Family Children's Hospital, Madison, Wisconsin, United States

REFERENCES:
- [Background] Mittal V. Family-centered rounds. Pediatr Clin North Am. 2014 Aug;61(4):663-70. doi: 10.1016/j.pcl.2014.04.003. PMID 25084715
- [Background] Seltz LB, Zimmer L, Ochoa-Nunez L, Rustici M, Bryant L, Fox D. Latino families' experiences with family-centered rounds at an academic children's hospital. Acad Pediatr. 2011 Sep-Oct;11(5):432-8. doi: 10.1016/j.acap.2011.06.002. Epub 2011 Jul 23. PMID 21783452
- [Background] COMMITTEE ON HOSPITAL CARE and INSTITUTE FOR PATIENT- AND FAMILY-CENTERED CARE. Patient- and family-centered care and the pediatrician's role. Pediatrics. 2012 Feb;129(2):394-404. doi: 10.1542/peds.2011-3084. Epub 2012 Jan 30. PMID 22291118
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Webster PD, Johnson BH. Developing Patient- and Family-Centered Vision, Mission, and Philosophy of Care Statements. Bethesda, MD: Institute of Family-Centered Care; 1999:55.
- [Background] Johnson B, Abraham M, Conway J, Simmons L, Edgman-Levitan S, Sodomka P, Schlucter J, Ford D. Partnering With Patients and Families to Design a Patient- and Family-Centered Health Care System: Recommendations and Promising Practices. Bethesda, MD: Institute for Patient- and Family-Centered Care; 2008.
- [Background] Davidson JE, Powers K, Hedayat KM, Tieszen M, Kon AA, Shepard E, Spuhler V, Todres ID, Levy M, Barr J, Ghandi R, Hirsch G, Armstrong D; American College of Critical Care Medicine Task Force 2004-2005, Society of Critical Care Medicine. Clinical practice guidelines for support of the family in the patient-centered intensive care unit: American College of Critical Care Medicine Task Force 2004-2005. Crit Care Med. 2007 Feb;35(2):605-22. doi: 10.1097/01.CCM.0000254067.14607.EB. PMID 17205007
- [Background] Mittal VS, Sigrest T, Ottolini MC, Rauch D, Lin H, Kit B, Landrigan CP, Flores G. Family-centered rounds on pediatric wards: a PRIS network survey of US and Canadian hospitalists. Pediatrics. 2010 Jul;126(1):37-43. doi: 10.1542/peds.2009-2364. Epub 2010 Jun 29. PMID 20587682
- [Background] Sisterhen LL, Blaszak RT, Woods MB, Smith CE. Defining family-centered rounds. Teach Learn Med. 2007 Summer;19(3):319-22. doi: 10.1080/10401330701366812. PMID 17594229
- [Background] Roter D, Larson S. The Roter interaction analysis system (RIAS): utility and flexibility for analysis of medical interactions. Patient Educ Couns. 2002 Apr;46(4):243-51. doi: 10.1016/s0738-3991(02)00012-5. PMID 11932123
- [Background] Roter DL, Larson S. The relationship between residents' and attending physicians' communication during primary care visits: an illustrative use of the Roter Interaction Analysis System. Health Commun. 2001;13(1):33-48. doi: 10.1207/S15327027HC1301_04. No abstract available. PMID 11370921
- [Background] Cooper LA, Roter DL, Johnson RL, Ford DE, Steinwachs DM, Powe NR. Patient-centered communication, ratings of care, and concordance of patient and physician race. Ann Intern Med. 2003 Dec 2;139(11):907-15. doi: 10.7326/0003-4819-139-11-200312020-00009. PMID 14644893
- [Background] Cox ED, Raaum SE. Discussion of alternatives, risks and benefits in pediatric acute care. Patient Educ Couns. 2008 Jul;72(1):122-9. doi: 10.1016/j.pec.2008.01.025. Epub 2008 Mar 17. PMID 18343624
- [Background] Cox ED, Smith MA, Brown RL. Evaluating deliberation in pediatric primary care. Pediatrics. 2007 Jul;120(1):e68-77. doi: 10.1542/peds.2006-2602. PMID 17606551
- [Background] Sorra JS, Dyer N. Multilevel psychometric properties of the AHRQ hospital survey on patient safety culture. BMC Health Serv Res. 2010 Jul 8;10:199. doi: 10.1186/1472-6963-10-199. PMID 20615247
- [Background] Cox ED, Smith MA, Brown RL, Fitzpatrick MA. Effect of gender and visit length on participation in pediatric visits. Patient Educ Couns. 2007 Mar;65(3):320-8. doi: 10.1016/j.pec.2006.08.013. Epub 2006 Oct 2. PMID 17011738
- [Background] Cypress BS. Family presence on rounds: a systematic review of literature. Dimens Crit Care Nurs. 2012 Jan-Feb;31(1):53-64. doi: 10.1097/DCC.0b013e31824246dd. PMID 22156815
- [Background] Tarini BA, Lozano P, Christakis DA. Afraid in the hospital: parental concern for errors during a child's hospitalization. J Hosp Med. 2009 Nov;4(9):521-7. doi: 10.1002/jhm.508. PMID 19653281
- [Result] Xie A, Carayon P, Cartmill R, Li Y, Cox ED, Plotkin JA, Kelly MM. Multi-stakeholder collaboration in the redesign of family-centered rounds process. Appl Ergon. 2015 Jan;46 Pt A:115-23. doi: 10.1016/j.apergo.2014.07.011. Epub 2014 Aug 12. PMID 25124394
- [Result] Xie A, Carayon P, Cox ED, Cartmill R, Li Y, Wetterneck TB, Kelly MM. Application of participatory ergonomics to the redesign of the family-centred rounds process. Ergonomics. 2015;58(10):1726-44. doi: 10.1080/00140139.2015.1029534. Epub 2015 Apr 22. PMID 25777042
- [Result] Kelly MM, Xie A, Carayon P, DuBenske LL, Ehlenbach ML, Cox ED. Strategies for improving family engagement during family-centered rounds. J Hosp Med. 2013 Apr;8(4):201-7. doi: 10.1002/jhm.2022. Epub 2013 Mar 6. PMID 23468375
- [Result] Carayon P, Li Y, Kelly MM, DuBenske LL, Xie A, McCabe B, Orne J, Cox ED. Stimulated recall methodology for assessing work system barriers and facilitators in family-centered rounds in a pediatric hospital. Appl Ergon. 2014 Nov;45(6):1540-6. doi: 10.1016/j.apergo.2014.05.001. Epub 2014 Jun 2. PMID 24894378
- [Result] Cox ED, Carayon P, Hansen KW, Rajamanickam VP, Brown RL, Rathouz PJ, DuBenske LL, Kelly MM, Buel LA. Parent perceptions of children's hospital safety climate. BMJ Qual Saf. 2013 Aug;22(8):664-71. doi: 10.1136/bmjqs-2012-001727. Epub 2013 Mar 29. PMID 23542553
- [Result] Benjamin JM, Cox ED, Trapskin PJ, Rajamanickam VP, Jorgenson RC, Weber HL, Pearson RE, Carayon P, Lubcke NL. Family-initiated dialogue about medications during family-centered rounds. Pediatrics. 2015 Jan;135(1):94-101. doi: 10.1542/peds.2013-3885. Epub 2014 Dec 15. PMID 25511116